CLINICAL TRIAL: NCT03769571
Title: Generalized Training Program for Caregivers on the ESDM
Brief Title: Generalized Training Program for Caregivers on the ESDM: PEGASE
Acronym: PEGASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-42
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parental coaching program at ESDM (P-ESDM) (Other)
  Interventions: Behavioral: Parental coaching program at ESDM (P-ESDM)
- CONTROL (No Intervention)

INTERVENTIONS:
Behavioral: Parental coaching program at ESDM (P-ESDM) — It will have a duration of 7 months (with an inclusion period of 1 year). Parents will come to the hospital with their child once every 15 days for one-hour parental coaching sessions on the ESDM method. Home video sessions will also be performed by parents once every 15 days. Each parent will have a Certified therapist referral to the practice of ESDM and the program is framed by a certified therapist and trained in ESDM parental coaching.
  Arms: parental coaching program at ESDM (P-ESDM)

SUMMARY:
The main objective of the study is to evaluate the effectiveness of a parent's training program (name PEGASE) of young children (aged 2 to 4 years) with Autism Spectrum Disorders.

This study is follow up by the Autism Resource Center PACA (CRA PACA), which is located in Marseille's university Department of Child Psychiatry.

This center is a regional expert center in diagnostic and research missions in the field of Autism. The center is promoting new advances in the field of Autism Spectrum Disorders (ASD) The center receives requests for diagnostic assessment from all the region. Autism is to date a major public health problem, current prevalence rates are 1 child / 88 in the United States. This prevalence continues to increase.

Autism is a severe neurodevelopment disorder with significant functional impact.

An essential axis in the field of health is to develop new treatment strategy including low costs and family impact particularly in quality of life.

In France, consensus guidelines (HAS 2012) on the diagnosis assessment for Autism Spectrum Disorders (ASD) people and interventions were edited.

Support for grade recommendations have been issued. In this research, the investigators focus on a global, early and coordinated management method: the Early Start Denver Model. This intervention obtained a grade B to the recommendations of the HAS in 2012. Early Start Denver Model (ESDM) is scientifically proven by a lots of studies.

Two management modalities are discuss in the ESDM model: the classical ESDM and the ESDM P (parents ESDM). Even if in both ways of care, the parent is put in a central position around the care of the child. In P ESDM, the parent is trained in the techniques of ESDM itself. This parental coaching program at ESDM (P-ESDM) was developed by Rogers et al at Sacramento Davis University.

P ESDM is not yet developed in France and has not been the subject of any French-language publication to date.

This program is dedicated to young parents of children with autism spectrum disorders aged between 2 and 4 years old.

This is a 7-month program (with a duration of inclusion of 3 year). The program is based on ESDM techniques, it meets both the need to include parents in care and the idea of reducing the cost of these care (need fewer hours of care by professionals).

This program is offered to all parents of autism spectrum disorders children between the ages of 2 and 4 who go to CRA PACA for an expert diagnostic evaluation.

The aim of this study is to objectify the effectiveness of this parental intervention in a French population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 4 years
* Child diagnosed with the clinical criteria of The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and International Classification of Diseases 10th Revision (ICD 10). Initial diagnosis of Autism spectrum disorder (ASD) should be validated by recommended diagnostic scales: ADI R, ADOS 2.
* A child whose parents or legal representatives have accepted their child's participation in this study, and have signed informed consent.

Exclusion Criteria:

* No presentation to initial and final evaluations
* Withdrawal of informed consent (which can intervene at any time of the study and without proof)

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-11-07 (Estimated); Study Completion 2021-11-07 (Estimated)

PRIMARY OUTCOMES:
effectiveness of a parent's training program (name PEGASE) of young children (aged 2 to 4 years) with Autism Spectrum Disorders. | 7 month
  Autism Diagnostic Observation Schedule 2 (ADOS 2) : Assessment of social affect and restricted and repetitive behaviours, autism severity level/Selected module
  The scale is between 0 and 3 :
  * Note 0 is assigned when the behavior does not show abnormalities specific to the disorders invasive development;
  * Note 1 is assigned when the behaviour is slightly abnormal or slightly unusual;
  * Note 2 corresponds to a clearly abnormal behaviour;
  * Note 3 is attributed to a frankly abnormal behavior, to the point that it interferes with the interaction. This note may also correspond to such a limited behaviour as the assessment of its quality social security is impossible.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier Arnaud, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de pédopsychiatrie Sainte-Marguerite, Marseille, Marseille Cedex 09, France